CLINICAL TRIAL: NCT03338946
Title: Evaluation of Cardiac Implanted Electronic Devices (CIED) "Readers" for Hospital Disease Management
Brief Title: Evaluation of CIED "Readers" for Disease Management
Status: Completed | Type: Observational
Sponsor: Edward Hospital (Other)
Responsible Party: Principal Investigator, Janet Gifford, Nurse Practitioner, Edward Hospital
Organization: Edward-Elmhurst Health System (Other)
Other Study IDs: Edward Hospital
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pacemaker Ddd; ICD
Keywords: Remote monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CIED subjects: CIED interrogation
  Interventions: Device: CIED interrogation

INTERVENTIONS:
Device: CIED interrogation — CareLink Express interrogation
  Other Names: Remote monitoring

SUMMARY:
The purpose of this study is to evaluate the use of remote interrogation (readers) of CIEDs in evaluation of suspected TIA/stroke patients, HF or those experiencing syncope. This approach has the potential to advance the practice of CIED evaluation by staff without specialized training in cardiac electrophysiology (non-EP staff). We hypothesize that actionable events will be identified with use of CIED readers. These events may include identification of atrial fibrillation in TIA/stroke patients, percentage biventricular pacing in patients with HF or evaluation of arrhythmic events in syncope patients. We believe that non-EP staff will find CIED readers easy or very easy to use and that time from transmission to analysis for non-EP trained staff will be low.

DETAILED DESCRIPTION:
Subjects with CIEDs undergoing evaluation for TIA/stroke, HF or syncope will be reviewed for inclusion/exclusion criteria. CIED interrogation, demographics and time of interrogation will be collected. Review of interrogation and medical record will be done to evaluate for actionable events including CIED programming, initiation or change in medications, admission/discharge or decision for further testing.

ELIGIBILITY:
Inclusion Criteria:

* have a Medtronic CIED compatible with Medtronic CareLink Express
* being evaluated for heart failure, TIA/stroke or syncope
* able to read and speak English

Exclusion Criteria:

-CIED from other than Medtronic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects being seen in Edward ED, HF clinic or inpatient units being evaluated for HF, TIA/stroke or syncope
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Incidence of actionable events after use of readers in suspected TIA/stroke, heart failure and syncope | one day
  percent of those with events after reader review with actions such as admission/discharge, addition or change in medications, further testing

SECONDARY OUTCOMES:
Average number of minutes from transmission to analysis | one day
  number of minutes from CareLink Express interrogation to analysis

OTHER OUTCOMES:
Incidence of non-EP trained staff rating CIED readers as very easy or easy | one year
  Likert scale to staff on ease of use

CONTACTS AND LOCATIONS:
Overall Officials: Janet Gifford, MSN, Principal Investigator — Edward Hospital
Locations (1):
- Edward Hospital, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided